CLINICAL TRIAL: NCT03053466
Title: A Phase 1 Multicenter, Dose Escalation, Cohort Extension and Dose and Disease Expansion Study of APL-501 in Subjects With Select Advanced or Relapsed/Recurrent Solid Tumors
Brief Title: APL-501 Study for Select Advanced or Relapsed/Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apollomics (Australia) Pty. Ltd. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry); Apollomics Inc. (formerly CBT Pharmaceuticals, Inc.) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-501-01
Record Dates: First submitted 2017-01-30; First posted 2017-02-15 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Solid Tumor; Microsatellite Instability; Mismatch Repair Deficiency; Cancer of Unknown Primary Site
Keywords: Advanced Solid Tumor; Relapsed Solid Tumor; Recurrent Solid Tumor
MeSH Terms: conditions — Microsatellite Instability; Turcot syndrome; Neoplasms, Unknown Primary

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm (Experimental): APL-501
  Interventions: Drug: APL-501

INTERVENTIONS:
Drug: APL-501 — Subjects will be assigned to a dose level in the order of study entry. Treatment includes a minimum of four 28-day cycles at three planned dose levels (1, 3, and 10 mg/kg). In the Dose Escalation Segment, each treatment cycle is comprised of 2 doses of study drug administered on Days 1 and 15 of a 28-day cycle. In the Cohort Extension, the treatment cycle will consist of 2 doses of study drug administered on Days 1 and 15 of a 28-day cycle.
  In Dose and Disease Expansion, the treatment cycle will consist of 2 doses of study drug (non-weight based dosing of 400 mg) administered on Days 1 and 15 of a 28-day cycle.
  Other Names: GB226; genolimzumab

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and recommended dose schedule of APL-501 in individuals with advanced or relapsed or recurrent solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, 3-part study with a Dose-Escalation Segment, Cohort Extension and Dose and Disease Expansion cohorts of APL-501 injection, a humanized IgG4 monoclonal antibody, targeting the Programmed Death-1 (PD-1) membrane receptor on T lymphocytes and other cells of the immune system. Select advanced solid tumor malignancies will receive escalating doses of APL-501.

Dose escalation will occur in three subject cohorts until a protocol defined dose limited toxicity (DLT) occurs, not due to disease progression or inter-current illness, and a tentative maximum tolerated dose (MTD) or biologically effective dose (BED) is determined.

Cohort Extension will evaluate APL-501 at 3 mg/kg and 10 mg/kg on Day 1 and Day 15 every 28 days.

At the tentative MTD, BED or recommended Phase 2 dose (RP2D), at least two tumor types in the Dose and Disease Expansion will be assessed at an equivalent non-weight based dose to further evaluate toxicity and preliminary efficacy.

ELIGIBILITY:
Major Inclusion Criteria:

• Able to understand and comply with study procedures, understand the risks involved, and provide written informed consent.

Dose Escalation:

* Histologically and / or cytological confirmed solid tumors: colorectal, endometrial, gastric including, gastroesophageal junction adenocarcinoma (GC), head and neck (esophageal, hepatocellular (HCC), non-small cell lung cancer, mesothelioma, ovarian, and renal cell carcinoma (RCC), either refractory or relapsed to standard therapy or for which no effective standard therapy is available.
* No restriction to number of prior therapies for Dose Escalation Segment except for gastric and renal cell carcinoma.

Cohort Extension:

* Histologically and/or cytological confirmed solid tumors with an approved labelled indication for PD-1 inhibitors.
* Tumor biopsy at study entry and during therapy. Tumor sites used to satisfy this criterion must not have received any prior radiation therapy. Sites for biopsy must be distinct from target lesions used for efficacy assessment.
* Measurable disease according to RECIST v1.1.

Dose and Disease Expansion:

* MSI-H or dMMR per local laboratory and failed at least one prior line of standard of care chemotherapy per local standards.
* Carcinoma of Unknown Primary

Major Exclusion Criteria:

* History of severe hypersensitivity to mAbs, excipients of the drug product or other components
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast
* Any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PDL-2, or anti-CTLA-4 antibody (or any other antibody targeting T cell co-stimulation pathways) (except NSCLC)
* Known significant mental illness or other conditions such as active alcohol or other substance abuse that, in the opinion of the Investigator, predisposes the subject to high risk of noncompliance with the protocol treatment or assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE v4.03) in patients with advance solid tumors | From the time of informed consent from signature until Day 28 after Cycle 1; Dose Escalation - Approximately 9 months
  Adverse events, serious adverse events, dose limiting toxicities according to the National Cancer Institute (NCI) Terminology Criteria for Adverse Events (CTCAE v4.03)

SECONDARY OUTCOMES:
Determine the recommended Phase 2 dose and schedule | An average of 1 year
  adverse events, serious adverse events, dose limiting toxicities
Area under the plasma concentration versus time curve (AUC) | Up to 4 months (1 cycle = 28 days)
  AUC, 0-infinity
Maximum plasma concentration | Up to 4 months (1 cycle = 28 days)
  Cmax
Time to reach Cmax | Up to 4 months (1 cycle = 28 days)
  Tmax
Objective Response Rate (ORR) | Approximately 24 months
  The treatment effect of APL-501 will be assessed by RECIST v1.1 and by irRECIST to determine proportion of patients with complete response or partial response.
Duration of Response (DOR) | Approximately 24 months
  The treatment effect of APL-501 will be assessed by RECIST v1.1 or by irRECIST to determine duration of response. Time from first documented complete response or partial response until subsequent documented disease progression or death.
Time to Response (TTR) | Approximately 24 months
  The treatment effect of APL-501 will be assessed by RECIST v1.1 and by irRECIST to determine time to complete response and partial response.
Disease Control Rate (DCR) | Approximately 24 months
  The treatment effect of APL-501 will be assessed by RECIST v1.1 and irRECIST to determine disease control rate. Proportion of patients with best overall response of complete response, partial response, or stable disease.
Progression Free Survival | Approximately 24 months
  The effect of APL-501 will be assessed by RECIST v1.1 and per irRECIST to determine progression free survival as time from date of first dose to date of disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Franco, Study Director — Apollomics Inc.
Locations (5):
- Australia (5):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Cabrini Health Limited, Malvern, Victoria
  - Peter MaCallum Cancer Centre, Melbourne, Victoria
  - Nucleus Network, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website for Apollomics Inc. — http://www.apollomicsinc.com/